CLINICAL TRIAL: NCT06594978
Title: Effects of Dual-site Anodal Transcranial Direct Current Stimulation on Attention, Decision-making and Working Memory During Sports Fatigue in Elite Soccer Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020070H
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sports Fatigue
Keywords: transcranial direct current stimulation; primary motor cortex; prefrontal cortex; cognitive function; sports fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dual-site anodal tDCS over the M1 (Experimental)
  Interventions: Device: dual-site anodal tDCS over the M1
- dual-site anodal tDCS over the DLPFC (Experimental)
  Interventions: Device: dual-site anodal tDCS over the DLPFC
- sham tDCS (Sham Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: dual-site anodal tDCS over the M1 — M1: motor cortex
  Arms: dual-site anodal tDCS over the M1
Device: dual-site anodal tDCS over the DLPFC — DLPFC: dorsolateral prefrontal cortex
  Arms: dual-site anodal tDCS over the DLPFC
Device: sham tDCS — sham stimulation
  Arms: sham tDCS

SUMMARY:
Investigation of the effects of dual-site anodal transcranial direct current stimulation over the dorsolateral prefrontal cortex or primary motor cortex on attention, decision-making and working memory during sports fatigue in elite soccer athletes

ELIGIBILITY:
Inclusion Criteria:

* elite soccer athletes

Exclusion Criteria:

* goalkeepers
* pregnancies
* family history of epilepsy
* metallic head implants
* neurological, psychiatric, or musculoskeletal disorders
* severe sports injuries

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Stroop task | immediately after the tDCS/sham-tDCS intervention
Reaction times of the Stroop task | immediately after the tDCS/sham-tDCS intervention
Net score in the Iowa Gambling task | immediately after the tDCS/sham-tDCS intervention
Hits in the 2-back task | immediately after the tDCS/sham-tDCS intervention
Misses in the 2-back task | immediately after the tDCS/sham-tDCS intervention
Reaction times in the 2-back task | immediately after the tDCS/sham-tDCS intervention
Index d' in the 2-back task | immediately after the tDCS/sham-tDCS intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sports, Exercise and Brain Sciences Laboratory, Sports Coaching College, Beijing Sport University, Beijing 100084, China, Beijing, Haidian, China

REFERENCES:
- [Derived] Qi F, Zhang N, Nitsche MA, Yi L, Zhang Y, Yue T. Effects of Dual-Site Anodal Transcranial Direct Current Stimulation on Attention, Decision-Making, and Working Memory during Sports Fatigue in Elite Soccer Athletes. J Integr Neurosci. 2025 Jan 21;24(1):26401. doi: 10.31083/JIN26401. PMID 39862014